CLINICAL TRIAL: NCT05627960
Title: FIH Phase 1A /1B Study of AG01 Antibody Against Progranulin/GP88 in Advanced Solid Tumor Malignancies With Expansion Cohorts in Advanced Triple Negative Breast Ca, Hormone Resistant Breast Ca, Non Small Cell Lung Cancer and Mesothelioma
Brief Title: First in Human Phase 1 Study of AG01 Anti-Progranulin/GP88 Antibody in Advanced Solid Tumor Malignancies
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: A&G Pharmaceutical Inc. (Industry)
Collaborators: University of Maryland Greenebaum Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GCC1950
Record Dates: First submitted 2022-03-16; First posted 2022-11-28 (Actual); Last update posted 2022-11-28 (Actual); Status verified 2022-11

CONDITIONS: Triple Negative Breast Cancer; Hormone-Resistant Breast Cancer; Non Small Cell Lung Cancer; Mesothelioma
Keywords: Progranulin; Advanced solid malignancies; Phase 1; Anti-Progranulin antibody; Advanced solid tumors; Breast Cancer; Lung Cancer; Mesothelioma
MeSH Terms: conditions — Triple Negative Breast Neoplasms; Carcinoma, Non-Small-Cell Lung; Mesothelioma; Breast Neoplasms; Lung Neoplasms | interventions — AG-01 compound

STUDY DESIGN:
Intervention Model Description: For dose escalation, model is an accelerated titration design-1-(3+3)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- AG-01 treated group phase 1A (Experimental): For dose escalation, subjects will be treated with increasing doses of AG01 from 1 mg/kg to 8 mg/kg. The duration of each treatment cycle is 28 days with two infusions of AG01 every 14 days.
  Interventions: Drug: AG-01 Compound
- AG-01 1B triple negative breast cancer treated group (Experimental): TNBC is defined as ER and/or PR < 1% by IHC, HER2 <3+ by IHC and/or FISH negative, subjects must have received 1 or more standard of care (SOC) therapies for metastatic TNBC.
  If PD(L)1-positive, must have received a combination of chemotherapy and a PD (L)-1 agent (Pembrolizumab), unless not a candidate for these therapies If gBRCA 1 or 2 mutation is present, must have received SOC therapies including a PARPi, unless not a candidate for these therapies.
  Sacituzumab Govitecan ADC is FDA approved for treatment of advanced TNBC, prior exposure to this therapy does not preclude eligibility in the current study.
  Interventions: Drug: AG-01 Compound
- AG-01 1B Hormone-resistant breast cancer (Experimental): Hormone-resistant breast cancer is defined as, ER and/or PR >1%, HER2 <3+ by IHC and/or FISH negative, received 1 or more hormonal (HT) therapies or HT/CD4/6 kinase inhibitor or HT/MTOR inhibitor for treatment of metastatic breast cancer. If the tumor has known PIK3CA mutation, HT/Alpelisib combination should be considered unless not a candidate for this therapy.
  Interventions: Drug: AG-01 Compound
- AG-01 1B NSCLC (Experimental): Subjects with metastatic/recurrent NSCLCA failed 2 or more SOC therapies, including platinum-based chemotherapy and an anti-PD (L) -1 agent (sequentially or consecutively), Subjects with sensitizing mutations/alterations/rearrangements are eligible if received 1 or more SOC agent/s targeting these mutations unless not a candidate for these therapies.
  Interventions: Drug: AG-01 Compound
- AG-01-1B mesothelioma (Experimental): Subjects with mesothelioma who received at least 1 SOC therapy for metastatic/recurrent mesothelioma per NCCN guidelines or not a candidate for SOC therapy.
  Interventions: Drug: AG-01 Compound

INTERVENTIONS:
Drug: AG-01 Compound — Phase 1A dose escalation study: enrolled subjects with advanced solid tumors will receive AG-01 compound at various doses.
  Phase 1B patients will be treated with AG-01 at the RP2D.

SUMMARY:
This is a first in human phase 1 study of AG01 an anti-Progranulin/Glycoprotein88 (PGRN/GP88) antibody in patients with advanced solid tumors. AG01 is a recombinant monoclonal antibody expressed in a CHO production cell line. The antibody AG01 binds to human PGRN/GP88, expressed on cancer cells.

This study will have a dose escalation portion (1A) to evaluate maximum tolerated dose (MTD) and/or maximum administered dose (MAD), the safety and tolerability of AG01treatment before the dose expansion portion (1B) of the study is initiated. The dose escalation portion of this study (1A) will also be used to determine the recommended phase 2 dose (RP2D) of AG01 antibody to be evaluated in the cohort expansion portion (1B).

DETAILED DESCRIPTION:
PGRN/GP88 is an 88 kilodalton glycoprotein produced by cells of epithelial or mesenchymal origin. It is an autocrine growth factor, which is overexpressed in several human cancers including breast and ovarian cancer, multiple myeloma, prostate cancer, non small cell as well as other tumors. High GP88 expression is associated with the malignant phenotype, increased proliferation and survival associated with drug resistance to some currently used therapeutic agents. Pathological studies have shown that PGRN/GP88 is an independent prognostic factor in several cancers including breast, non-small cell lung carcinoma, prostate and digestive cancers. High GP88 expression in tumor tissues is associated with decreased disease-free survival and increased mortality. In addition, in stage 4 breast cancer patients, high circulating level of PGRN/GP88 is associated with decreased overall survival.

This study will enroll patients with relapsed/refractory solid tumor malignancies (1A) who failed one or more standard chemotherapy or targeted therapy regimens per SOC guidelines such as NCCN guidelines and for whom no standard therapy exists. In 1B portion of the study patients with triple negative breast cancer, hormone resistant breast cancer, non small cell lung cancer and mesothelioma will be accrued. The treatment period (cycle) will consist of 28-day cycles, the AGO1 will be infused every 14 days. The dosing schedule/frequency of treatments for subjects in the dose escalation portion (1A) will be the same as for subjects in the expansion portion (1B).

ELIGIBILITY:
Inclusion Criteria:

1. Signed informed consent/authorization is obtained prior to conducting any study-specific screening procedures.
2. 18 years of age or older.
3. Histologic or cytologic diagnosis of advanced cancer.
4. Radiographic evidence of at least 1 measurable metastatic lesion per RECIST 1.1 criteria.
5. Patients with relapsed/refractory solid tumor malignancies who failed one or more standard chemotherapy or targeted therapy regimens per SOC guidelines such as NCCN guidelines and for whom no standard therapy exists (Phase 1A). No GP88 expression pre-required for phase 1A.
6. For phase 1B, patients must have GP88 tissue tumor tissue expression of 1+, 2+ or 3+ by IHC, archival tumor tissue will be used whenever possible. If no archival tissue is available, subject will be asked to consent to a study specific tumor biopsy for GP88 testing (phase1B). Patients who do not have archival tissue available for the dose expansion cohort (1B) will not be exposed to significant risk procedure to obtain tissue and may still be eligible for the study, after discussion with the Sponsor and Medical Monitor.
7. At least 4 weeks after the last dose of chemotherapy or radiation therapy; 6 weeks for mitoxantrone or mitomycin therapy.
8. ECOG performance status must be ≤2 (Appendix A).
9. Adequate hepatic, renal, and bone marrow function:

   Absolute neutrophil count ≥ 1,000/uL Platelets ≥ 100,000/µL Total bilirubin WNL per Institution ULN AST (SGOT)/ALT (SGPT) ≤ 2.5 X institutional ULN Creatinine ≤1.2 mg/dL Clearance ≥50ml/min (Cockcroft-Gault)
10. All study participants (male and female) with reproductive potential must practice highly effective methods of contraception (failure rate <1% annually) while on this study and for 90 days after completion of study therapy.
11. Men and women of all ethnic groups are eligible for this trial.
12. Females at reproductive age must have a negative urine pregnancy test prior to entry to this study.
13. Males with partners at reproductive age must use highly effective birth control methods to prevent partners' pregnancy while on study and for 90 days after completion of study treatments.
14. Life expectancy is greater than 12 weeks.
15. Subjects with triple negative breast cancer (TNBC) cohort must have received 1 or more standard of care (SOC) or targeted therapies for metastatic TNBC. If PD(L)1-positive, must have received a combination of chemotherapy and a PD (L)-1 agent (Atezolizumab or Pembrolizumab), unless not a candidate for these therapies. If gBRCA 1 or 2 mutation is present, must have received SOC therapies including a PARPi, unless not a candidate for these therapies. is FDA approved for treatment of advanced TNBC. Prior exposure to Sacituzumab Govitecan ADC therapy does not preclude eligibility in the current study.
16. Subjects with Cohort 2-Breast Cancer ER and/or PR positive, hormone-resistant breast cancer who received 1 or more hormonal (HT) therapies or HT/CD4/6 kinase inhibitor or HT/MTOR inhibitor for treatment of metastatic breast cancer are eligible. If the tumor has known PIK3CA mutation, HT/Alpelisib combination should be considered unless not a candidate for this therapy.
17. Subjects with metastatic/recurrent NSCLCA who failed 2 or more SOC therapies, including platinum-based chemotherapy and an anti-PD (L) -1 agent (sequentially or consecutively). Patients with sensitizing mutations/alterations/rearrangements are eligible if received 1 or more SOC agent/s targeting these mutations unless not a candidate for these therapies.
18. Mesothelioma patients who have received at least 1 SOC therapy for metastatic/recurrent mesothelioma per NCCN recommendations or not a candidate for SOC therapy.

Exclusion Criteria:

1. Uncontrolled inter-current illness including, but not limited to, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmias not well controlled with medication, myocardial infarction within the previous 6 months, or psychiatric illness/social situations that would limit compliance with study requirements.
2. Uncontrolled or untreated CNS metastases and treated CNS metastases are allowed, as long as the patient is clinically stable.
3. Presence carcinomatous meningeal involvement.
4. Patients may not be receiving any other investigational agents, or have participated in any investigational drug study < 28 days prior to starting on the current study.
5. Since the teratogenic potential of AG01 is currently unknown, females who are pregnant or lactating are excluded.
6. Males and females unable to adhere to abstinence or use highly effective methods of contraception (annual failure rate < 1%) to prevent study subjects' pregnancy or study subjects' partner pregnancy.
7. History of any other malignancies in the last 2 years except for in-situ cancer, basal or squamous cell skin cancer treated with curative intent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 77 (Estimated)
Dates: Start 2022-02-14 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-11 (Estimated)

PRIMARY OUTCOMES:
Maximum Tolerated Dose (MTD) and/or Maximum Administered Dose (MAD) | 28 days during 1st cycle
  Determine the MTD and/or MAD of anti GP88 monoclonal antibody (AG-01) in subjects with advanced/refractory solid tumor malignancies for which no effective therapies exist.
Antitumor Activity of AG-01 by Overall Response Rate (ORR) | Every 56 Days
  To evaluate the antitumor activity of AG-01 monoclonal antibody as assessed by ORR defined as complete response (CR), partial response (PR), stable disease >24 weeks (SD) (CR+PR+ SD) based on RECIST v1.1 in subjects with TNBC, ER+ hormone resistant Breast Cancer, NSCLCA and mesothelioma.
  Each cohort will be assessed separately for response.

SECONDARY OUTCOMES:
Recommended phase 2 dose (RP2D) of AG-01-Phase 1A | 28 days or 1cycle
  During 1A portion accelerated titration (1pt/dose) design will be utilized to guide dose progression and estimation of the maximum tolerated dose MTD and/or maximum administered dose (MAD) (1). Once treatment related DLT occurs, this cohort will be expanded to 3+3 design, and all subsequent cohorts will follow the 3+3 design.
  First dose/cohort level subjects will be monitored for 28 days from the D1 of the 1st infusion of AG01 (2 doses, D 1 and D15 of AG01) before the dose is escalated to the next dose level without expansion of cohort and assuming no DLTs during this time.
Safety and tolerability of AG-01 | While receiving AG-01 for 56 days and for 30 days after the last dose of the study drug (day 86)
  Subjects will be monitored for emergence of any adverse events; with physical exams, laboratory assessments, ECOG PS, Vital signs, changes in weight, clinical symptoms. Adverse events will be assessed via CTACE V 5.0 on ongoing basis in Phase 1A and 1B:
Pharmacokinetic (PK) profile of AG-01-1A | Day 1 (cycle1 first dose), Day 4, Day 8, Day 15 (cycle 1 second dose), day 29 (Cycle 2 first dose), day 43 (cycle 2 second dose), Day 46, Day 50, Day 57 (end of treatment) and Day 87 (30 days post end of treatment).
  Blood samples will be collected collected in cycles 1 and 2, End of Treatment and 30 days post-treatment, per study schedule to determine AG01 drug levels and PK profile.
Preliminary anti-tumor activity of the AG-01 in subjects with refractory/advanced solid tumor malignancies (1A and 1B). | While receiving AG-01 treatment, at day 56
  Response to treatment with AG-01 will be assessed with tumor imaging (CTs/MRIs/Bone scan-as applicable) every 56 days, response will be assessed via RECIST 1.1
Anti-drug antibodies (ADA) to AG-01 | Day 1 (cycle1 first dose) Day 15 (cycle 1 second dose), day 29 (Cycle 2 first dose), day 43 (cycle 2 second dose), Day 57 (end of treatment),and Day 87 (30 days post end of treatment)
  ADA blood samples will be collected prior to AG-01 administration on Days 1, 15, 29, and 43 with blood sampling following the described time frame and tested via immunoassay for presence anti-AG01 antibodies

OTHER OUTCOMES:
Serial Glycoprotein88 (GP-88) blood levels | Day 1 (cycle1 first dose) Day 15 (cycle 1 second dose), day 29 (Cycle 2 first dose), day 43 (cycle 2 second dose), Day 57 (end of treatment),and Day 87 (30 days post end of treatment).
  Exploratory outcome-To determine the serial GP88 blood levels using the available ELISA blood test while on treatment with the Anti-GP88 monoclonal antibody (AG01).

CONTACTS AND LOCATIONS:
Overall Officials: Katherine Tkaczuk, MD, Principal Investigator — University of Maryland, Baltimore
Locations (1):
- University of Maryland Greenebaum Comprehensive Cancer Center, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Serrero G. Potential of Theranostic Target Mining in the Development of Novel Diagnostic and Therapeutic Products in Oncology: Progranulin/GP88 as a Therapeutic and Diagnostic Target for Breast and Lung Cancers. Rinsho Byori. 2016 Nov;64(11):1296-1309. PMID 30695312
- [Background] Tkaczuk KHR, Hawkins D, Yue B, Hicks D, Tait N, Serrero G. Association of Serum Progranulin Levels With Disease Progression, Therapy Response and Survival in Patients With Metastatic Breast Cancer. Clin Breast Cancer. 2020 Jun;20(3):220-227. doi: 10.1016/j.clbc.2019.11.010. Epub 2019 Dec 5. PMID 31928925
- [Background] Koo DH, Do IG, Oh S, Lee YG, Kim K, Sohn JH, Park SK, Yang HJ, Jung YS, Park DI, Jeong KU, Kim HO, Kim H, Serrero G, Chun HK; KBSMC Colorectal Cancer Team. Prognostic Value of Progranulin in Patients with Colorectal Cancer Treated with Curative Resection. Pathol Oncol Res. 2020 Jan;26(1):397-404. doi: 10.1007/s12253-018-0520-7. Epub 2018 Oct 30. PMID 30378010
- [Background] Greither T, Steiner T, Bache M, Serrero G, Otto S, Taubert H, Eckert AW, Kappler M. GP88/PGRN Serum Levels Are Associated with Prognosis for Oral Squamous Cell Carcinoma Patients. Biology (Basel). 2021 May 4;10(5):400. doi: 10.3390/biology10050400. PMID 34064411
- [Background] Guha R, Yue B, Dong J, Banerjee A, Serrero G. Anti-progranulin/GP88 antibody AG01 inhibits triple negative breast cancer cell proliferation and migration. Breast Cancer Res Treat. 2021 Apr;186(3):637-653. doi: 10.1007/s10549-021-06120-y. Epub 2021 Feb 22. PMID 33616772
- [Background] Serrero G, Hawkins DM, Bejarano PA, Ioffe O, Tkaczuk KR, Elliott RE, Head JF, Phillips J, Godwin AK, Weaver J, Hicks D, Yue B. Determination of GP88 (progranulin) expression in breast tumor biopsies improves the risk predictive value of the Nottingham Prognostic Index. Diagn Pathol. 2016 Aug 8;11(1):71. doi: 10.1186/s13000-016-0520-4. PMID 27501955
- [Background] Edelman MJ, Feliciano J, Yue B, Bejarano P, Ioffe O, Reisman D, Hawkins D, Gai Q, Hicks D, Serrero G. GP88 (progranulin): a novel tissue and circulating biomarker for non-small cell lung carcinoma. Hum Pathol. 2014 Sep;45(9):1893-9. doi: 10.1016/j.humpath.2014.05.011. Epub 2014 Jun 5. PMID 25033727
- [Background] Serrero G, Hawkins DM, Yue B, Ioffe O, Bejarano P, Phillips JT, Head JF, Elliott RL, Tkaczuk KR, Godwin AK, Weaver J, Kim WE. Progranulin (GP88) tumor tissue expression is associated with increased risk of recurrence in breast cancer patients diagnosed with estrogen receptor positive invasive ductal carcinoma. Breast Cancer Res. 2012 Feb 8;14(1):R26. doi: 10.1186/bcr3111. PMID 22316048
- [Background] Arechavaleta-Velasco F, Perez-Juarez CE, Gerton GL, Diaz-Cueto L. Progranulin and its biological effects in cancer. Med Oncol. 2017 Nov 7;34(12):194. doi: 10.1007/s12032-017-1054-7. PMID 29116422
- [Background] Abrhale T, Brodie A, Sabnis G, Macedo L, Tian C, Yue B, Serrero G. GP88 (PC-Cell Derived Growth Factor, progranulin) stimulates proliferation and confers letrozole resistance to aromatase overexpressing breast cancer cells. BMC Cancer. 2011 Jun 9;11:231. doi: 10.1186/1471-2407-11-231. PMID 21658239
- [Background] Wong NC, Cheung PF, Yip CW, Chan KF, Ng IO, Fan ST, Cheung ST. Antibody against granulin-epithelin precursor sensitizes hepatocellular carcinoma to chemotherapeutic agents. Mol Cancer Ther. 2014 Dec;13(12):3001-12. doi: 10.1158/1535-7163.MCT-14-0012. Epub 2014 Sep 24. PMID 25253787